CLINICAL TRIAL: NCT05492396
Title: Evaluation of Healing Following Open Gluteus Medius Repair Augmented With a Biointegrative Implant
Brief Title: Evaluation of Healing Following Open Gluteus Medius Repair With Biointegrative Implant
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, William Vasileff, Associate Professor, Ohio State University
Other Study IDs: 2021H0451
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hip Injuries; Tendon Injuries; Orthopedic Procedures
MeSH Terms: conditions — Hip Injuries; Tendon Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Standard gluteus medius repair: Subjects will all undergo standard gluteus medius repair that includes augmentation with the biointegrative implant.
  Interventions: Device: Standard gluteus medius repair with Tapestry Biointegrative implant

INTERVENTIONS:
Device: Standard gluteus medius repair with Tapestry Biointegrative implant — Patients will undergo standard gluteus medius repair utilizing augmentation.

SUMMARY:
This is a prospective, single-center study design with enrollment of 15 subjects. The 15 subjects will all undergo standard gluteus medius repair that includes augmentation with the biointegrative implant. This is a small observational study. As such, we expect that the results from 15 subjects will give an adequate understanding of post surgical healing.

DETAILED DESCRIPTION:
Surgical gluteal tendon repair is a procedure performed regularly in operating rooms everywhere. This procedure is normally recommended to address gluteal tendon tears after nonoperative treatment options have been exhausted. However, less than satisfactory long-term outcomes can be common after open gluteal tendon repair. The augmentation of tendon repairs via various biointegrative implants is becoming more common in clinical practice, however very little, if any, of the literature details the healing after surgical intervention.

Biointegrative implants have been studied for the use of augmenting other tendon repairs, such as rotator cuff tears. Successful complete rotator cuff repairs augmented with a collagen-based implant have indicated that biointegrative implants are a safe option that may provide greater rates of healing and more positive long-term outcomes (Thon SG, 2019). Rates of healing and long-term outcomes when using a patch of this sort in other tendons such as the gluteal tendon in the hip show promise and demonstrate that there is a need for this area of study.

A 2016 study evaluated augmenting gluteus medius repair with a bioinductive implant, but the surgery was performed using endoscopic technique. There is no literature studying the healing of collagen-based implants for open gluteal tendon repairs. Although clinical outcomes show similar level of improvement for endoscopic and open gluteal tendon tear repair (Maslaris A, 2020), open repair technique with more anchors may be required for larger or more intricate tears.

This is a prospective, single-center study design with enrollment of 15 subjects. The 15 subjects will all undergo standard gluteus medius repair that includes augmentation with the biointegrative implant. This is a small observational study. As such, we expect that the results from 15 subjects will give an adequate understanding of post surgical healing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years of age
2. Patients healthy enough to undergo procedure
3. Large partial tear and full thickness gluteal tendon tear requiring augmentation
4. Willing and able to make all required visits
5. Able to read and write in English

Exclusion Criteria:

1. Hypersensitivity or objection to using bovine derived materials
2. Significant atrophy or major retraction of gluteal tendon
3. Women who are pregnant or nursing
4. History of poor compliance with medical treatment
5. Patients who are incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a gluteal tendon tear where surgical repair is indicated will be screened for inclusion. Those that meet all inclusion criteria and no exclusion criteria will be invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Assess overall tissue quality by ultrasound assessment | 6 month
  Graded as 'Intact/Attenuated/Disrupted'. Intact being the positive outcome, disrupted being the negative outcome.
Assess overall tissue thickness by ultrasound assessment | 6 month
  Unit measured in centimeters
Assess overall tissue organization by ultrasound assessment | 6 month
  Hypoechoic signal present or absent. Present being the positive outcome, absent being the negative outcome

SECONDARY OUTCOMES:
Modified Harris Hip Score questionnaire | Screening, 6 weeks, 3 month, 6 month, 12 months
  Measures the functional status of the hip. Scores range from 0-100 where 100 means best functional outcome and least pain
International Hip Outcome Tool questionnaire | Screening, 6 weeks, 3 month, 6 month, 12 months
  Assesses deficiencies with respect to outcome assessment of patients with hip disorders. Scores range from 0-100. Higher scores represent better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: William K Vasileff, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Jameson Crane Sports Medicine Institute, Columbus, Ohio
  - The Ohio State University Hospital East, Columbus, Ohio
  - Ohio State Outpatient Care New Albany, Westerville, Ohio

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared